CLINICAL TRIAL: NCT07248787
Title: Effect of Multi-Sensory Interventions Applied to Pregnant Women on Labor Pain, Comfort, and Satisfaction
Brief Title: Effect of Multi-Sensory Interventions on Labor Pain, Comfort, and Birth Satisfaction
Acronym: MSI-LABOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Fatma Aybice Karaca, Midwife, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaU-EBE-MSI-RCT-2025
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Labor Pain; Birth Satisfaction
Keywords: Labor pain; Aromatherapy; Massage therapy; Music therapy; Visual stimulation; Comfort; Birth satisfaction; Multi-sensory intervention; Midwifery; Supportive care
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Five parallel groups: sacral massage, lavender aromatherapy, Turkish makam music, aquarium visual stimulus, and control (standard care).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and statisticians will be blinded to group assignments during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sacral Massage (Experimental): Participants in this group will receive a 10-minute sacral massage during each stage of labor (three times in total) by a trained midwife using circular hand movements over the sacral area to relieve labor pain.
  Interventions: Behavioral: Sacral Massage
- Lavender Aromatherapy (Experimental): Participants in this group will receive lavender aromatherapy through a diffuser for 20 minutes during each stage of labor (three times in total). A few drops of pure lavender essential oil will be added to distilled water in a diffuser to promote relaxation and reduce pain perception.
  Interventions: Behavioral: Lavender Aromatherapy
- Turkish Makam Music (Experimental): Participants will listen to selected Turkish Makam music (Rehavi and Nihavend) played at 45-65 dB for 20 minutes during each stage of labor (three times in total). Music will be delivered via headphones in a quiet environment to enhance comfort and emotional well-being.
  Interventions: Behavioral: Turkish Makam Music
- Aquarium Visual Stimulus (Experimental): Participants will watch a video of an aquarium scene (fish swimming calmly) displayed on a screen throughout the active phase of labor to provide a soothing visual focus and reduce anxiety.
  Interventions: Behavioral: Aquarium Visual Stimulus
- Standard Care (No Intervention): Participants in the control group will receive routine obstetric care without any additional sensory interventions.

INTERVENTIONS:
Behavioral: Sacral Massage — A 10-minute sacral massage applied by a trained midwife during each stage of labor (three sessions in total). The massage involves circular hand motions to relieve pain and promote relaxation.
  Arms: Sacral Massage
Behavioral: Lavender Aromatherapy — Lavender essential oil diffused for 20 minutes during each stage of labor (three times total) to promote calmness and reduce pain intensity.
  Arms: Lavender Aromatherapy
Behavioral: Turkish Makam Music — Rehavi and Nihavend Turkish makam music (45-65 dB) played through headphones for 20 minutes during each stage of labor (three times total).
  Arms: Turkish Makam Music
Behavioral: Aquarium Visual Stimulus — Continuous presentation of an aquarium scene video during the active phase of labor to provide visual distraction and relaxation.
  Arms: Aquarium Visual Stimulus

SUMMARY:
The goal of this clinical trial is to learn whether different multi-sensory methods can help lower labor pain and improve comfort and birth satisfaction among pregnant women giving birth vaginally.

The main questions this study aims to answer are:

Do supportive methods such as massage, lavender aromatherapy, Turkish makam music, or aquarium visual stimulation help women feel less labor pain compared to standard care?

Do these methods increase women's comfort and satisfaction during labor?

Participants will be randomly assigned to one of five groups:

Sacral massage group - will receive 10-minute sacral massages three times during labor.

Lavender aromatherapy group - will inhale lavender essential oil through a diffuser for 20 minutes, three times during labor.

Music therapy group - will listen to Turkish makam music (Rehavi or Nihavend) for 20 minutes, three times during labor.

Visual stimulation group - will watch a live aquarium image continuously during active labor.

Control group - will receive standard maternity care only.

All participants will give informed consent and receive care in the obstetrics unit of Kütahya City Hospital, Türkiye.

Researchers will measure:

Labor pain intensity at 4-5 cm, 6-7 cm, and 8-10 cm cervical dilatation using a Visual Analogue Scale (VAS).

Comfort level at 8-9 cm using the Comfort Characteristics Questionnaire (CCQ).

Birth satisfaction about 2 hours after delivery using the Birth Satisfaction Scale (BSS).

Labor duration will also be recorded.

This study will help determine which sensory methods are most effective and comfortable for pregnant women, and may guide supportive care practices during childbirth.

DETAILED DESCRIPTION:
This study investigates the effects of four non-pharmacological, multi-sensory interventions-sacral massage, lavender aromatherapy, Turkish makam music, and aquarium visual stimulation-on key intrapartum outcomes. The trial uses a five-arm, parallel-group, randomized design conducted in the obstetrics clinic of Kütahya City Hospital.

Participants will be randomly assigned using sealed, opaque envelopes. All sensory interventions will be applied during the active and transitional phases of labor by trained midwives following standardized procedures. Outcome assessment will be performed by personnel blinded to group allocation to minimize bias.

The rationale for the selected sensory interventions is based on their proposed ability to modulate pain perception, enhance relaxation, and support emotional well-being through tactile, olfactory, auditory, or visual pathways. Each method has been previously used in maternity care, though comparative evidence in a multi-arm design is limited.

The study will evaluate the safety, feasibility, and relative effectiveness of these interventions within routine clinical practice. Analyses will follow the intention-to-treat principle. Standard comparative tests (e.g., ANOVA and repeated-measures models) will be used to examine differences in pain trajectories and other outcomes across the five groups.

The findings aim to generate clinically relevant evidence supporting the integration of culturally appropriate sensory strategies into intrapartum care to enhance women's childbirth experiences.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 to 40 years
* Gestational age ≥ 37 weeks (term pregnancy)
* Singleton pregnancy with cephalic presentation
* Expected vaginal delivery
* Cervical dilation of at least 3 cm at hospital admission
* Able to communicate in Turkish and provide informed consent

Exclusion Criteria:

* Diagnosed high-risk pregnancy (e.g., preeclampsia, placenta previa, fetal distress)
* History of cesarean section or uterine surgery
* Use of epidural, spinal anesthesia, or opioid analgesics during labor
* Visual, auditory, or olfactory impairments that may affect perception of the interventions
* Allergy or sensitivity to lavender oil
* Emergency cesarean section or any complication requiring medical intervention
* Refusal or withdrawal of consent at any stage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Labor Pain Level | Assessed at 4-5 cm, 6-7 cm, and 8-10 cm cervical dilation during active labor.
  Pain intensity measured using a 10-cm VAS at three points in active labor.

SECONDARY OUTCOMES:
Comfort Level (Comfort Scale) | At 8-9 cm cervical dilation during active labor
  Maternal comfort during labor will be measured using the Comfort Scale developed by Kolcaba.
Birth Satisfaction (Birth Satisfaction Scale) | Up to 2 hours postpartum.
  Maternal satisfaction with the childbirth experience will be evaluated using the Birth Satisfaction Scale (BSS) approximately 2 hours after delivery. Higher scores indicate greater satisfaction.
Labor Duration | From 3 cm cervical dilation until delivery (up to approximately 12-18 hours).
  Total duration of labor (minutes) will be calculated as the time from 3 cm cervical dilation to delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya City Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.